CLINICAL TRIAL: NCT03311542
Title: Expanded Access for Pembrolizumab (MK-3475) to Patients With Melanoma or Glioblastoma / Glioma After Failed Standart Therapy, at High Mutational Load Which is Confirmed by the Results of Molecular-genetic Analysis of Tumor Tissue.
Brief Title: Expanded Access for Pembrolizumab (MK-3475)
Status: No longer available | Type: Expanded Access
Sponsor: Center Trials & Treatment (Other)
Responsible Party: Sponsor
Other Study IDs: PST-2-B
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Melanoma (Skin); Melanoma Recurrent; Glioblastoma Multiforme; Glioblastoma by Gene Expression Profile; Glioma of Brain
Keywords: GBM; Glioma
MeSH Terms: conditions — Melanoma; Glioblastoma; Glioma | interventions — pembrolizumab

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: pembrolizumab — Each participant will receive pembrolizumab every 21 days for up to 12 month or until confirmed disease progression on MRI or CT, unacceptable toxicity, confirmed.positive pregnancy test or withdrawal of consent.
  Other Names: MK-3475

SUMMARY:
This is an expanded access program (EAP) for patient with Melanoma and Glioblastoma who have progressed after prior Protocol therapy including Bevacizumab, Temozolomide ( TMZ ), Ipilimumab, BRAF and MEK inhibitors. The patients whose tumors are EGFR, MET or ALK positive should first receive an EFGR or ALK inhibitor, respectively, prior to treatment with pembrolizumab.

DETAILED DESCRIPTION:
Pembrolizumab has been approved by the U.S. Food and Drug Administration for the treatment of patients with Glioblastoma and Melanoma The Expanded Access Program (EAP) for this medicine in the U.S. is closed. The EAP will continue outside the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Patient's willing to sign Informed Consent.
* Unresectable metastatic Melanoma / Glioblastoma / Glioma.
* Failed or progressed on standard of care systemic therapy including bevacizumab, ipilimumab, radiotherapy, regardless of prior treatment with a BRAF/ MEK/ EGFR/ MET/ ALK inhibitors, as long as all other eligibility criteria for this study are met.
* Female participants of childbearing potential must be willing to use adequate contraception or be surgically sterile, or abstain from heterosexual activity starting with the first dose of treatment through at least 120 days after the last dose of pembrolizumab.
* Male participants must agree to use an adequate method of contraception starting with the first dose of treatment through 120 days after the last dose of pembrolizumab.
* Results of partial genomic or full-genomic sequencing or genetic studies to determine the status of the patient's mutation load.
* ECOG performance status greater than or equal to 2
* Adequate kidney function: serum creatinine less than or equal to 2.0 mg/dL or creatinine clearance greater than or equal to 40 mL/min
* Adequate bone marrow function: absolute neutrophil count greater than or equal to 1.5 x 10^9/L, hemoglobin greater than or equal to 10 g/dL (can be corrected by growth factor or transfusion), and platelet count greater than or equal to 100 x 10^9/L
* Adequate liver function: total bilirubin less than or equal to 1.5 x upper limit of normal (ULN), alkaline phosphatase, alanine aminotransferase, and aspartate aminotransferase less than or equal to 3 x ULN (or less than or equal to 5 x ULN in case of liver metastases). If alkaline phosphatase is greater than 3 x ULN (in absence of liver metastases) or greater than 5 x ULN (in presence of liver metastases) AND patient also is known to have bone metastases, the liver specific alkaline phosphatase must be used to assess liver function instead of total alkaline phosphatase
* Willing and able to comply with all aspects of the treatment protocol

Exclusion Criteria:

* Eligibility for any other pembrolizumab study open in the same region.
* Existing anti-cancer therapy-related toxicities of grade 2 or more, except that alopecia and grade 2 neuropathy are acceptable.
* History of congestive heart failure with New York Heart Association Classification greater than grade II, unstable angina, myocardial infarction within the past 6 months or serious cardiac arrhythmia.
* Electrocardiogram with QTc interval of greater than or equal to 500 msec based upon Bazett's formula (QTcB).
* The Investigator believes the patient to be medically unfit to receive pembrolizumab or unsuitable for any other reason.
* Pregnancy (positive B-hCG test) or breastfeeding.
* Hypersensitivity to pembrolizumab.
* Use of corticosteroids for this indication has been discontinued for at least 4 weeks before starting treatment in this protocol.
* History of or concomitant medical condition that, in the opinion of the Investigator, would compromise the patient's ability to safely complete the treatment protocol.
* Meningeal carcinomatosis.
* Pulmonary lymphangitic involvement resulting in pulmonary dysfunction requiring active treatment, including use of oxygen.
* Not recovered from minor or major surgery and less than 4 weeks from major surgery
* History of life-threatening or severe immune-related adverse events on treatment with another immunotherapy.
* Expected to require any other form of systemic antineoplastic therapy while receiving pembrolizumab.
* History of clinically severe autoimmune disease (e.g., requires chronic immunosuppressive therapy).
* History of pneumonitis, organ transplant, human immunodeficiency virus (HIV), active hepatitis B or hepatitis C.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- N.N. Alexandrov National Cancer Centre, Minsk, Belarus
- The Hong Kong Cancer Institute, Hong Kong, Hong Kong
- "Cancer Research Center" of the Ministry of Health of the Republic of Tajikistan, Dushanbe, Tajikistan
- Republican Cancer Research Center of the Ministry of Health of the Republic of Uzbekistan (RENTC MH RUz), Tashkent, Uzbekistan

REFERENCES:
- [Background] Kottschade LA, McWilliams RR, Markovic SN, Block MS, Villasboas Bisneto J, Pham AQ, Esplin BL, Dronca RS. The use of pembrolizumab for the treatment of metastatic uveal melanoma. Melanoma Res. 2016 Jun;26(3):300-3. doi: 10.1097/CMR.0000000000000242. PMID 26848796
- [Background] Buiar PG, de Azevedo SJ. Atypical Presentation: Metastatic Uveal Melanoma in a Young Patient without Visual Complaints. Front Oncol. 2017 May 18;7:99. doi: 10.3389/fonc.2017.00099. eCollection 2017. PMID 28573105
- [Background] Preusser M, Lim M, Hafler DA, Reardon DA, Sampson JH. Prospects of immune checkpoint modulators in the treatment of glioblastoma. Nat Rev Neurol. 2015 Sep;11(9):504-14. doi: 10.1038/nrneurol.2015.139. Epub 2015 Aug 11. PMID 26260659